CLINICAL TRIAL: NCT03214601
Title: A Prospective, Multicenter, Non-Blinded, Non-Randomized Early Feasibility Study of the Relay Branch Thoracic Stent-Graft System in Subjects With Thoracic Aortic Pathologies Requiring Treatment Proximal to the Origin of the Innominate Artery
Brief Title: Early Feasibility Study of the RelayBranch Thoracic Stent-Graft System
Acronym: RelayBranch
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0019-16
Record Dates: First submitted 2017-06-25; First posted 2017-07-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Thoracic Aorta Aneurysm; Aneurysm, Ruptured; Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aneurysm, Ruptured; Aortic Aneurysm | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: The Relay Branch System is intended for treating thoracic aortic arch pathologies requiring coverage of the innominate and left common carotid arteries. The system includes a graft with a proximal landing zone in the proximal aorta and branch grafts that extend into the innominate and left common carotid arteries. The arch graft and branch grafts are composed of self-expanding nitinol stents sutured to polyester vascular graft fabric, creating an exoskeleton
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Relay Branch System (Experimental): Subjects who receive the Relay Branch System for repair which includes those with aneurysmal disease, penetrating atherosclerotic ulcer (PAU), and chronic uncomplicated Type B aortic dissection.
  Interventions: Device: penetrating atherosclerotic ulcer, aorta branch cardiovascular implant

INTERVENTIONS:
Device: penetrating atherosclerotic ulcer, aorta branch cardiovascular implant — The Relay Branch System is intended to provide an option for patients with arch and proximal descending chronic thoracic aortic pathologies.
  Other Names: Relay Branch System; system, endovascular graft, aortic aneurysm treatment

SUMMARY:
The purpose of this study is to conduct an early clinical evaluation of the Relay Branch System, which will provide initial insight into the clinical safety and function of the device.

This Early Feasibility Study (EFS) will assess the safety and effectiveness of the device at the index procedure and at 30-day follow-up. The study will evaluate the delivery and deployment of the device, patency of branches and branch vessels, and exclusion of the aortic pathology. The data will help determine if modifications need to be made to the device, the procedural steps, operator technique, or the indications for use.

DETAILED DESCRIPTION:
This Early Feasibility Study (EFS) protocol describes the clinical study requirements for the Relay Branch System; a device designed to provide an option for patients with arch and proximal descending chronic thoracic aortic pathologies. As an EFS, this investigation is intended to provide proof of principle and initial clinical safety data on the Relay Branch System. The study is planned as an initial investigation of the device for aortic arch and proximal descending thoracic aortic aneurysmal disease, PAU (including IMH) and uncomplicated chronic Type B aortic dissection (including IMH). The study will yield information on procedural techniques; assessing the safety and effectiveness of the device at the index procedure and at 30 days, focusing on device delivery and deployment, and circulatory exclusion of the pathologic process. As a branched device, patency of the endograft branches will also be assessed.

The study will evaluate three-dimensional (3D) imaging data, both at baseline and through follow-up. Baseline 3D anatomy will augment information on the precise anatomic configuration of patients presenting aortic arch pathology treatable with the device. Follow-up imaging will provide information on the effectiveness of the device with respect to endoleaks in patients with aneurysms, sealing of dissections, PAU and IMH, and stability of the device at the deployed position, response, endograft patency, and short-term device integrity.

The data from this EFS will yield insights into the following aspects of the device, preceding a traditional feasibility or pivotal study:

* The clinical safety of the device-specific aspects of the procedure,
* Determination of delivery and deployment of the device,
* Operator-dependent aspects of device use,
* Human factors associated with the design and use of the device,
* Safety of the device as assessed by device-related adverse events,
* Effectiveness of the device in performing its intended purpose over short-term follow-up.

Observations from the study will guide the instructions for use (IFU) for the device. Finally, the study will collect imaging data to augment the current use conditions data set. It is anticipated that information collected will be used to make applicable design changes, or be combined with a prospective, investigational device exemption (IDE) study for submission of an original premarket approval application (PMA) to the U.S. Food and Drug Administration (FDA) for approval to commercially distribute the system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Anatomy that would require coverage of the brachiocephalic trunk (BCT) and/or left carotid arteries if a non-branch endograft were implanted
* At least one of the following:

  a. Aneurysm of the ascending aorta, aortic arch, or proximal descending aorta that meets at least one of the following: i. ≥ 5.5 cm in diameter ii. ≥ 4.0 cm in diameter that has increased in size by 0.5 cm in the last 6 months iii. Measures twice the size of the normal aorta diameter iv. Is saccular in configuration

  b. PAU within the ascending aorta, aortic arch, or proximal descending thoracic aorta (DTA) with or without intramural hematoma (IMH)

  c. Chronic, uncomplicated aortic dissection distal to the BCT (type B), with either aortic diameter ≥5.5 cm or ≥4.0 cm with an increase in size by 0.5 cm in the last 6 months d. IMH distal to the BCT with recurrent symptoms, i.e. hypertension or intractable pain, despite best medical therapy.
* A non-aneurysmal proximal aortic neck diameter ranging between 28 mm and 43 mm and a non-aneurysmal distal aortic neck diameter ranging between 19 mm and 43 mm.
* A proximal attachment zone of the arch graft, meeting the oversizing requirement, must be a minimum of 25mm in length when measured on the inner curve of the ascending aorta, proximal to the BCT.
* Total length from the coronaries to the proximal edge of the BCT must be a minimum of 70mm.
* The length of the distal landing zone should be 20mm minimum.
* Coverage of the left subclavian artery is permitted. Revascularization of the left subclavian artery may be considered in all cases by the treating physician and, especially, in anatomies where revascularization is determined to be clinically necessary
* The distal landing zone must contain a straight segment (non-tapered, non-reverse tapered; defined by < 10% diameter change) with length equal to or greater than the required attachment length of the intended device
* Non-aneurysmal BCT and left common carotid arteries with diameters ranging > 6.0mm across the entire length of the treatment zone.
* Distal branch landing zone must be <20.0 mm in diameter and a minimum of 25.0 mm in length.
* Adequate arterial access for introduction and delivery of the Relay Branch System. Note: Alternative methods to gain proper access can be utilized (e.g., iliac conduit)
* Considered high risk or prohibitive risk for conventional surgery by treating physician or aortic team
* Must be willing to comply with the follow-up evaluation schedule
* Subject or legally authorized representative must sign the informed consent form prior to implant.

Exclusion Criteria:

* Significant stenosis, calcification, thrombus, or tortuosity of intended fixation sites that would compromise fixation or seal of the device
* Aortic angulations (radius) less than 15mm at intended proximal landing zone.
* Ascending aortas that would require the arch graft to be deployed less than 15mm distal to the coronaries
* Pre-procedure occlusion or planned coverage of both subclavian arteries
* Anatomic variants which would compromise circulation to both vertebral arteries after placement of the stent-graft
* Prior endovascular repair in the ascending/descending thoracic aorta or aortic arch. The device may not be placed within any prior endovascular graft
* Concomitant aneurysm/disease of the abdominal aorta requiring repair
* Prior abdominal aortic aneurysm repair (endovascular or surgical) that was performed less than 6 months prior to the planned stent implant procedure
* Prior mechanical aortic valve replacement except for hybrid valves with biological leaflets.
* Major surgical or medical procedure within 45 days prior to the planned procedure or is scheduled for a major surgical or medical procedure within 60 days post implantation. Except for any planned procedures for the prospective stent-graft placement, e.g., left subclavian artery bypass or transposition
* Untreatable allergy or sensitivity to contrast media or device components
* Blood coagulation disorder or bleeding diathesis in which the treatment cannot be suspended for one week pre and post repair
* Acute Coronary Syndrome (ACS) including unstable angina
* Severe Congestive Heart Failure (New York Heart Association functional class IV)
* Stroke within 12 months of the planned treatment date
* Myocardial infarction within 3 months of the planned treatment date.
* Chronic atrial fibrillation or other hypercoagulable condition that requires treatment with anticoagulants or presence of left atrial appendage thrombus
* Severe pulmonary disease (documented FEVI <30% or as assessed by the study physician) at screening
* Acute renal failure (defined as serum creatinine > 2.5mg/dL Note: Patients that have chronic renal failure and are managed medically or through hemodialysis, and can tolerate the follow-up imaging schedule can be included.
* Significant carotid bifurcation disease (>70% diameter reduction by duplex ultrasound or angiography)
* Hemodynamic instability
* Active systemic infection at the time of treatment
* Morbid obesity or other condition that may compromise or prevent the necessary imaging requirements
* Connective tissue disorders, mycotic aneurysms, or infected aorta
* Less than two-year life expectancy
* Current or planned participation in an investigational drug or device study that has not completed primary endpoint evaluation
* Currently pregnant or planning to become pregnant during the course of the study
* Medical, social, or psychological issues that the Investigator believes may interfere with treatment or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Major Adverse Events (MAEs) | 30 days after the index procedure
  The primary safety outcome determined by the rate of MAEs, including
  * All-cause mortality
  * Disabling stroke: a Modified Rankin Score (mRS) of 2 or more at 90 days and an increase in at least one mRS category from an individual's pre-stroke baseline
  * Permanent Paralysis/Paraparesis
  * Spontaneous Myocardial Infarction according to the SCAI definition
  * Renal Failure
  * Procedural Blood Loss >1,000mL

SECONDARY OUTCOMES:
Composite of the following Criteria | Technical success will be evaluated in 2 stages; the first evaluation occurs during the implant procedure. Technical success is then re-evaluated again 30 days post operation to ensure the graft placement was successful as outlined above
  * Acute technical success evaluation, beginning with the insertion of the introducer sheath and as a composite of the following:
    1. Success is defined as a successful delivery of the device through (i.e. ability to deliver the implant to the intended implantation site, without the need for unanticipated corrective intervention related to delivery):
    2. Successful deployment of the device as defined as
    i. Deployment of the endovascular stent-graft at the intended implantation site; ii. Patency (<50%) of all components of the implant with absence of device deformations requiring unplanned placement of an additional device within the endovascular stent-graft; and iii. absence of inadvertent covering of aortic branch vessels; and
    c. Successful withdrawal of the delivery system
  * Patency of all endograft components at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Luis Sanchez, MD, Principal Investigator — Barnes Jewish Hospital, Washington Univ; Wilson Szeto, MD, Principal Investigator — Penn Presbyterian Medical Center
Locations (12):
- United States (12):
  - University of Southern California, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barnes Jewish Hospital at Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania/Penn Presbyterian, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Baylor Scott and White Research Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No